CLINICAL TRIAL: NCT05940805
Title: A Randomized Controlled Trial to Evaluate a Comprehensive Protocol With Four Therapeutic Modalities for the Treatment of Upper Limb Spasticity in Post-stroke Hemiplegic Patients
Brief Title: Comprehensive Protocol for Treatment of Upper Limb Spasticity in Post-stroke Hemiplegic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Wu Tu Hsing, Director of Center of Acupuncture of Orthopaedics and Traumatology Institute, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3853051109
Record Dates: First submitted 2023-06-06; First posted 2023-07-11 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Post-stroke Upper Limb Spasticity
Keywords: Muscle Spasticity; Stroke; Stroke Rehabilitation; Nerve Block; Dry Needling; Transcranial Direct Current Stimulation; Electric Stimulation Therapy
MeSH Terms: conditions — Muscle Spasticity; Stroke

STUDY DESIGN:
Intervention Model Description: Thirty-two subjects diagnosed with a stroke at least six months prior to the study were randomized to receive ten sessions of either the treatment protocol or a sham intervention. The treatment protocol consisted of transcranial low-frequency electrical stimulation using subcutaneous needles over the scalp, paraspinous blocks, spastic muscle needling and functional electrical stimulation. Spasticity, range of motion, pain, functionality and quality of life were evaluated.
Who Masked: Participant, Outcomes Assessor
Masking Description: The Sham Group received the four modalities of the intervention, but these modalities were all inactive. For simulation of transcranial electrical stimulation and FES, electrodes were placed on the scalp and in the upper extremity muscles and were connected to a device similar to the real electric current generator. This device did not transmit any electric current but had blinking lights and produced sound to provide the subjects visual and auditory feedback. To simulate dry needling and paraspinous block, retractile needles were used. The patients were blinded to their assigned treatment group. Blinded examiners evaluated patients at baseline, one week post-treatment and three months post-treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protocol Group (PG) (Experimental): The PG received the following combination of four therapeutic modalities twice a week for five weeks:
  1. Low-frequency transcranial electrical stimulation;
  2. Paraspinous block;
  3. Dry needling of spastic upper limb muscles;
  4. Muscular functional electrical stimulation (FES).
  Interventions: Procedure: Low-frequency transcranial electrical stimulation; Paraspinous block; Dry needling of spastic upper limb muscles; Muscular functional electrical stimulation (FES)
- Sham Group (SG) (Sham Comparator): The Sham Group also received the four modalities of the intervention, but these modalities were all inactive. For simulation of transcranial electrical stimulation and FES, electrodes were placed on the scalp and in the upper extremity muscles and were connected to a device similar to the real electric current generator. This device did not transmit any electric current but had blinking lights and produced sound to provide the subjects visual and auditory feedback. To simulate dry needling and paraspinous block, retractile needles were used. The patients were blinded to their assigned treatment group.
  Interventions: Procedure: SHAM Low-frequency transcranial electrical stimulation; Paraspinous block; Dry needling of spastic upper limb muscles; Muscular functional electrical stimulation (FES)

INTERVENTIONS:
Procedure: Low-frequency transcranial electrical stimulation; Paraspinous block; Dry needling of spastic upper limb muscles; Muscular functional electrical stimulation (FES) — 1. Low-frequency transcranial electrical stimulation (2/100 Hz) applied through 0.3-mm-diameter and 40-mm-long needles placed subcutaneously on the scalp at the projection of Penfield's motor homunculus and sensory and frontal supplementary motor associative areas.
  2. Paraspinous block at the levels of the C5, C6 and C7 vertebrae concordant with spasticity laterality.
  3. Dry needling of spastic upper limb muscles, as identified through a thorough physical examination, using 0.3-mm-diameter and 40-mm-long needles.
  4. Muscular functional electrical stimulation (FES) in the antagonists of the upper limb muscles with spasticity with the following parameters: 20-Hz frequency, 300-µs pulse width, zero-second ramp time, 5-second stimulation time, and 5-second resting time.
  Arms: Protocol Group (PG)
Procedure: SHAM Low-frequency transcranial electrical stimulation; Paraspinous block; Dry needling of spastic upper limb muscles; Muscular functional electrical stimulation (FES) — For simulation of transcranial electrical stimulation and FES, electrodes were placed on the scalp and in the upper extremity muscles and were connected to a device similar to the real electric current generator. This device did not transmit any electric current but had blinking lights and produced sound to provide the subjects visual and auditory feedback. To simulate dry needling and paraspinous block, retractile needles were used.
  Arms: Sham Group (SG)

SUMMARY:
The general objective of this study was to evaluate the efficacy of the comprehensive protocol in improving post-stroke upper limb spasticity. The specific objectives were to evaluate pain improvement and changes in quality of life and functional capacity in patients who were subjected to the comprehensive protocol compared with those in the patients who underwent sham interventions.

DETAILED DESCRIPTION:
Background: Managing post-stroke upper limb spasticity is a major challenge in the rehabilitation field. The objective of this study was to evaluate the efficacy of a comprehensive treatment protocol with four therapeutic modalities in the recovery of patients with chronic stroke by evaluating clinical, neurological and functional outcomes.

Methodology: Thirty-two subjects diagnosed with a stroke at least six months prior to the study were randomized to receive ten sessions of either the treatment protocol or a sham intervention. The treatment protocol consisted of transcranial low-frequency electrical stimulation using subcutaneous needles over the scalp, paraspinous blocks, spastic muscle needling and functional electrical stimulation. Spasticity, range of motion, pain, functionality and quality of life were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years;
* Diagnosis of ischemic or hemorrhagic stroke at least six months previously;
* Presence of single upper limb spasticity

Exclusion Criteria:

* Spasticity due to conditions other than stroke;
* Hypersensitivity to lidocaine;
* Use of cardiac pacemakers;
* Presence of coagulation disturbances;
* Insufficient perceptual and cognitive capacity to understand the proposed treatment and answer the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2023-11-12 (Actual); Study Completion 2023-12-03 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth scale | 3 months
  To measure spasticity, and shoulder, elbow and wrist active and passive goniometry was performed to measure range of motion improvement. Minimum value = 0 (No increase in tone); Maximum value = 4 (Affected part in rigid flexion and extension)
Visual analogue scale (VAS) | 3 months
  To measure patients pain after the interventions. Minimun value = 0 (Painless); Maximum value = 10 (painful)
Functional independence measure (FIM) | 3 months
  To measure independence of patients after the interventions. The Functional Independence Measure (FIM) is a functional assessment with 18 items in the areas of personal care, sphincter control, mobility, communication and social-cognition, through a broad questionnaire. Minimun value = 18 (total dependence); maximum value = 126 (total independence)
Quality of Life - SF-36 questionnaire | 3 months
  To measure patients' quality of life after the interventions for each domain. Minimum value (for each domain) = 0 (bad quality of life); Maximum value for each domain = 100 (good quality of life)

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo General Hospital, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Treger I, Shames J, Giaquinto S, Ring H. Return to work in stroke patients. Disabil Rehabil. 2007 Sep 15;29(17):1397-403. doi: 10.1080/09638280701314923. PMID 17729085
- [Background] Ovbiagele B, Nguyen-Huynh MN. Stroke epidemiology: advancing our understanding of disease mechanism and therapy. Neurotherapeutics. 2011 Jul;8(3):319-29. doi: 10.1007/s13311-011-0053-1. PMID 21691873
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Soliman EZ, Sorlie PD, Sotoodehnia N, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2012 update: a report from the American Heart Association. Circulation. 2012 Jan 3;125(1):188-97. doi: 10.1161/CIR.0b013e3182456d46. No abstract available. PMID 22215894
- [Background] Ones K, Yilmaz E, Cetinkaya B, Caglar N. Quality of life for patients poststroke and the factors affecting it. J Stroke Cerebrovasc Dis. 2005 Nov-Dec;14(6):261-6. doi: 10.1016/j.jstrokecerebrovasdis.2005.07.003. PMID 17904035
- [Background] Burke D, Wissel J, Donnan GA. Pathophysiology of spasticity in stroke. Neurology. 2013 Jan 15;80(3 Suppl 2):S20-6. doi: 10.1212/WNL.0b013e31827624a7. PMID 23319482
- [Background] Sunnerhagen KS, Olver J, Francisco GE. Assessing and treating functional impairment in poststroke spasticity. Neurology. 2013 Jan 15;80(3 Suppl 2):S35-44. doi: 10.1212/WNL.0b013e3182764aa2. PMID 23319484
- [Background] Schlaug G, Renga V, Nair D. Transcranial direct current stimulation in stroke recovery. Arch Neurol. 2008 Dec;65(12):1571-6. doi: 10.1001/archneur.65.12.1571. PMID 19064743
- [Background] Bhakta BB. Management of spasticity in stroke. Br Med Bull. 2000;56(2):476-85. doi: 10.1258/0007142001903111. PMID 11092096
- [Background] Gerwin RD. Myofascial pain and fibromyalgia: Diagnosis and treatment. J Back Musculoskelet Rehabil. 1998 Jan 1;11(3):175-81. doi: 10.3233/BMR-1998-11304. PMID 24572598
- [Background] Teasell RW, Foley NC, Bhogal SK, Speechley MR. An evidence-based review of stroke rehabilitation. Top Stroke Rehabil. 2003 Spring;10(1):29-58. doi: 10.1310/8YNA-1YHK-YMHB-XTE1. PMID 12970830
- [Background] Raju RS, Sarma PS, Pandian JD. Psychosocial problems, quality of life, and functional independence among Indian stroke survivors. Stroke. 2010 Dec;41(12):2932-7. doi: 10.1161/STROKEAHA.110.596817. Epub 2010 Oct 21. PMID 20966411
- [Background] Boyaci A, Topuz O, Alkan H, Ozgen M, Sarsan A, Yildiz N, Ardic F. Comparison of the effectiveness of active and passive neuromuscular electrical stimulation of hemiplegic upper extremities: a randomized, controlled trial. Int J Rehabil Res. 2013 Dec;36(4):315-22. doi: 10.1097/MRR.0b013e328360e541. PMID 23579106
- [Background] de Kroon JR, IJzerman MJ. Electrical stimulation of the upper extremity in stroke: cyclic versus EMG-triggered stimulation. Clin Rehabil. 2008 Aug;22(8):690-7. doi: 10.1177/0269215508088984. PMID 18678569
- [Background] Hara Y, Ogawa S, Muraoka Y. Hybrid power-assisted functional electrical stimulation to improve hemiparetic upper-extremity function. Am J Phys Med Rehabil. 2006 Dec;85(12):977-85. doi: 10.1097/01.phm.0000247853.61055.f8. PMID 17117002
- [Background] Wu D, Qian L, Zorowitz RD, Zhang L, Qu Y, Yuan Y. Effects on decreasing upper-limb poststroke muscle tone using transcranial direct current stimulation: a randomized sham-controlled study. Arch Phys Med Rehabil. 2013 Jan;94(1):1-8. doi: 10.1016/j.apmr.2012.07.022. Epub 2012 Aug 7. PMID 22878231
- [Background] Hara Y, Ogawa S, Tsujiuchi K, Muraoka Y. A home-based rehabilitation program for the hemiplegic upper extremity by power-assisted functional electrical stimulation. Disabil Rehabil. 2008;30(4):296-304. doi: 10.1080/09638280701265539. PMID 17852312
- [Background] Sahin N, Ugurlu H, Albayrak I. The efficacy of electrical stimulation in reducing the post-stroke spasticity: a randomized controlled study. Disabil Rehabil. 2012;34(2):151-6. doi: 10.3109/09638288.2011.593679. Epub 2011 Oct 15. PMID 21999668
- [Background] Ring H, Weingarden H. Neuromodulation by functional electrical stimulation (FES) of limb paralysis after stroke. Acta Neurochir Suppl. 2007;97(Pt 1):375-80. doi: 10.1007/978-3-211-33079-1_49. PMID 17691399
- [Background] Popovic DB, Popovic MB, Sinkjaer T. Neurorehabilitation of upper extremities in humans with sensory-motor impairment. Neuromodulation. 2002 Jan;5(1):54-66. doi: 10.1046/j.1525-1403.2002._2009.x. PMID 22151782
- [Background] Bergfeldt U, Skold C, Julin P. Short Form 36 assessed health-related quality of life after focal spasticity therapy. J Rehabil Med. 2009 Mar;41(4):279-81. doi: 10.2340/16501977-0318. PMID 19247549
- [Background] Childers MK, Brashear A, Jozefczyk P, Reding M, Alexander D, Good D, Walcott JM, Jenkins SW, Turkel C, Molloy PT. Dose-dependent response to intramuscular botulinum toxin type A for upper-limb spasticity in patients after a stroke. Arch Phys Med Rehabil. 2004 Jul;85(7):1063-9. doi: 10.1016/j.apmr.2003.10.015. PMID 15241751
- [Background] Kaptchuk TJ, Goldman P, Stone DA, Stason WB. Do medical devices have enhanced placebo effects? J Clin Epidemiol. 2000 Aug;53(8):786-92. doi: 10.1016/s0895-4356(00)00206-7. PMID 10942860
- [Background] Ratmansky M, Defrin R, Soroker N. A randomized controlled study of segmental neuromyotherapy for post-stroke hemiplegic shoulder pain. J Rehabil Med. 2012 Oct;44(10):830-6. doi: 10.2340/16501977-1021. PMID 22949162
- [Background] Cournan M. Use of the functional independence measure for outcomes measurement in acute inpatient rehabilitation. Rehabil Nurs. 2011 May-Jun;36(3):111-7. doi: 10.1002/j.2048-7940.2011.tb00075.x. PMID 21675396
- See also: Projeto Diretrizes da Associação Médica Brasileira e Conselho Federal de Medicina - Diagnóstico e Tratamento da Espasticidade. 2001. — http://www.projetodiretrizes.org.br/projeto_diretrizes/048.pdf